CLINICAL TRIAL: NCT06476535
Title: Observatory of Patients With MyeloProliferative Neoplasm Treated With Anti-inflammatory Immunotherapy
Acronym: OPIUM
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0155 - OPIUM
Record Dates: First submitted 2024-06-13; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Myeloproliferative Neoplasm; Inflammatory Disease
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will collect cases of MPN patients who also benefit from an anti-inflammatory immunotherapy for another disease. Efficacy and tolerability of the drug will be assessed in this population.

ELIGIBILITY:
Inclusion Criteria:

* MyeloProliferative Neoplasm diagnosis
* receiving or having received an immunotherapy targeting IL-1, IL-6, IL-17, IL-23 or TNF

Exclusion Criteria:

* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MyeloProliferative Neoplasm patients followed in one of the centres participating to the FIM (French Intergroup- MPN) group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the anti-inflammatory immunotherapy | 1 year
  Depending on the indication of the anti-inflammatory treatment, clinical efficacy will be assessed clinically as number of patients reaching complete (total disappearance of initial symptoms- diarrhea, arthritis, fever, skin lesions), partial (improvement of symptoms, but not total disappearance) or absence of response (the treatment did not improve the symptoms). Clinical judgement will be according to the physician appreciation.
Tolerability of the anti-inflammatory immunotherapy | 1 year
  Tolerability will be assessed as the number of reported unexpected side effects attributed to the treatment as judged by the caring physician, including treatment discontinuation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement